CLINICAL TRIAL: NCT04382469
Title: Egyptian Initial Experience About 2019 Novel Corona Virus Disease (COVID-19): Single-center Study Analysis of 48 Patients in Alexandria-Egypt Regarding Radiological Patterns and Co-morbid Lung Diseases
Brief Title: Egyptian Initial Experience About 2019 Novel Corona Virus: Study of 48 Patients in Alexandria-Egypt Using Chest CT
Status: Completed | Type: Observational
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Ahmed Samir, Lecturer of radio-diagnosis, Alexandria University
Other Study IDs: IRB (00012098), FWA (00018699)
Record Dates: First submitted 2020-05-05; First posted 2020-05-11 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: COVID

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Corona virus disease 2019 (COVID-19) is a highly infectious disease caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).

Purpose: To give initial experience about COVID-19 in Alexandria-Egypt describing radiological patterns of lung involvement, also surveying prevalence of co-morbid lung diseases and their effect on COVID-19 presentation.

Methods: Retrospective study including 48 patients with positive polymerase chain reaction (PCR) test for COVID-19 during the period from February 2020 till May 2020 in Alexandria/Egypt. Full clinical and laboratory data are obtained. High resolution computed tomography (HRCT) findings are described. Serial follow up studies are done. Surveying co-morbid lung diseases done including tuberculosis (TB), interstitial lung diseases (ILDs), chronic obstructive lung disease (COPD), immune and vascular-related diseases. Prevalence rate is the predominant analysis.

DETAILED DESCRIPTION:
1. Study population and medical records review:

   * This retrospective study in Alexandria/Egypt during the period from February 2020 till May 2020, approved by out Institutional Ethics Committee. Patient consent waived by the Research Ethics Board, assuring respect of patient and medical records confidentiality. No overlap with any previously published work.
   * Forty-eight Egyptian patients with proved COVID-19 test results to be enrolled in this study without age or sex limitations.
   * Complete medical records to be obtained including thorough history taking and clinical examination. This include patient age and sex, smoking history, exposure history (including direct contact to positive COVID-19 patient or recent travelling to high risk countries¬, also health care providers to positive COVID-19 patients).
   * Present history to be taken regarding patient chest or general complaint.
   * Past history to be acquired regarding general chronic or debilitating diseases and cardio-pulmonary co-morbid diseases including TB, ILDs, COPD, immune and vascular related diseases.
   * Thorough general and local chest examination to be carried out.
   * Initial lab investigations to be obtained including complete blood count (CBC) and C-reactive protein) CRP. Blood gases and O2 saturation to be also reported.
   * Strict protocol of infection control to be followed during clinical assessment, laboratory work and radiological examinations according to the national and the international guidelines.
   * Exclusion criteria were: Incomplete medical records, degrade CT images because of patient tachypnea and motions artifacts, also unremarkable CT scans.
2. Clinical and laboratory data analysis:

   • The clinical and laboratory data to be obtained and analyzed by four consultant pulmonogists and single consultant chest pediatrician (having long time experience in clinical practice of chest infectious diseases and ICU patients for 20 to 33 years)
3. CT scanning and parameters:

   * CT examinations using multiple MDCT machines including Philips Brilliant-16, Siemens Emotion-64, Toshiba Aquilion-16, Toshiba Aquilion-64 and Toshiba Aquilion CXL/CX 128.
   * CT Scanning parameters: Slice thickness: 1 - 1.25 mm. Volumetric HRCT table speed that yields least cycles of breath holds as possible. Tube rotation: 0.6-0.9 second. Detector Collimation 1 mm. Helical mode (volumetric HRCT). kVp and mA per slice: 120 - 130 KVp and 200-400 mA, according to type of MSCT machine used, weight of the patient and clinical indication.
   * Positive intra-venous contrast administration only when prescribed.
4. CT analysis:

   • CT images to be viewed by four consultant radiologists (having long time experience in thoracic imaging ranging from 11 to 25 years) using either specialized work stations or Di-com viewers on personal computers with analysis of the axial, sagittal and coronal planes. MIP and Min-IP reconstructions to be routinely analyzed.
5. Statistical analysis:

Prevalence of clinico-laboratory data and HRCT findings estimated as the percentage of patients showing each criteria or abnormality.

ELIGIBILITY:
Inclusion Criteria:

* Positive COVID-19

Exclusion Criteria:

* Incomplete medical records, degrade CT images because of patient tachypnea and motions artifacts, also unremarkable CT scans.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Primary care centers
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Radiological pattern of initial presentation, disease progress, healing and recovery | "through study completion, an average of 1 month"
  HRCT findings
Survey of co-morbid lung diseases | "through study completion, an average of 1 month"
  prevalence

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Samir, MD, Principal Investigator — Department of Radio-diagnosis.
Locations (1):
- Faculty of Medicine, University of Alexandria, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No
The investigators will recommend further large group future researches for some notices in the study, but preferably not be biased